CLINICAL TRIAL: NCT01449435
Title: Asthma Exacerbations in Young Children With Moderate Asthma - Prospective Evaluation of Predictors
Brief Title: Predictors of Asthma Exacerbations in Children
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Cosultant Pediatric Allergy and Pulmonolgy, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU-238/11
Record Dates: First submitted 2011-10-07; First posted 2011-10-10 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Asthma
Keywords: Asthma; children; predictors of exacerbation; Methacholine challenge; Pulmonary function testing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Methacholine challenge testing — Nebulized methacholine administered at the following doses: 0,1 mg/0,4 mg/0,8 mg/1,6 mg
  Other Names: Aerosol Provocation System (Cardinal Health GmbH)

SUMMARY:
The purpose of this study is to determine whether parameters of the pulmonary function tests and the bronchial hyperresponsiveness to methacholine are predictors of asthma exacerbations.

DETAILED DESCRIPTION:
Preliminary investigations from our own research group showed that lung function parameters (FEV1, the FEV1/FVC ratio and a moderate to severe hyperresponsiveness to methacholine challenge were risk factors of asthma exacerbations (OR 11.3). In the present study, these parameters will be evaluated in prospective design.

One hundred children will be included in the study. Baseline parameters will be collected in a healthy interval (visit 1), then the children will be followed up for 1 year. If the patients fulfill the criteria for an exacerbation the children will present in our department. We expect that 44% of the children have an exacerbation. All children will present at a second visit after one year (visit 2).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >3 and <7 years
* Diagnosis of intermittent asthma
* In the last 24 months, at least 6 weeks of treatment with a controller medication (inhaled steroid and / or leukotriene receptor antagonist Singulair ®), or in the last 12 months, at least three episodes with an use of controller medications (inhaled steroid and / or the leukotriene receptor antagonist Singulair ®)
* The ability to perform three reproducible spirometries
* Examination in infection-free interval (> 4 weeks infection-free)
* Minimum distance to the following asthma medications:
* Short-acting beta 2-agonists: 8 hours
* Ipratropium bromide: 24 hours
* Long-acting beta 2-agonists: 24 hours
* steroids: 4 weeks
* leukotriene antagonist: 4 weeks

Exclusion Criteria:

* Age older than 6 years or younger than 4
* The inability to perform spirometry
* Other chronic diseases or infections (eg. HIV, tuberculosis, malignancy)
* Participation in another study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Outpatients of departement of Pediatric Pulmonology and Allergology.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | 1 year
  An exacerbations is defined as an increased need of salbutamol (more than two puffs per week or more than five puffs per two weeks). In this case patients will be followed up at our hospital and will start an anti-inflammatory therapy, if it is necessary.

SECONDARY OUTCOMES:
Predictors of exacerbations like lung function, nonspecific bronchial hyperresponsiveness to methacholine, exhaled NO, specific IgE, total IgE und ECP | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Background] Carlsen KH. What distinguishes the asthmatic amongst the infant wheezers? Pediatr Allergy Immunol. 1997;8(10 Suppl):40-5. No abstract available. PMID 9455779
- [Background] Castro-Rodriguez JA, Holberg CJ, Wright AL, Martinez FD. A clinical index to define risk of asthma in young children with recurrent wheezing. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1403-6. doi: 10.1164/ajrccm.162.4.9912111. PMID 11029352
- [Background] Kurukulaaratchy RJ, Matthews S, Holgate ST, Arshad SH. Predicting persistent disease among children who wheeze during early life. Eur Respir J. 2003 Nov;22(5):767-71. doi: 10.1183/09031936.03.00005903. PMID 14621083
- [Background] Kurukulaaratchy RJ, Matthews S, Arshad SH. Relationship between childhood atopy and wheeze: what mediates wheezing in atopic phenotypes? Ann Allergy Asthma Immunol. 2006 Jul;97(1):84-91. doi: 10.1016/S1081-1206(10)61375-0. PMID 16892787
- [Background] Thumerelle C, Deschildre A, Bouquillon C, Santos C, Sardet A, Scalbert M, Delbecque L, Debray P, Dewilde A, Turck D, Leclerc F. Role of viruses and atypical bacteria in exacerbations of asthma in hospitalized children: a prospective study in the Nord-Pas de Calais region (France). Pediatr Pulmonol. 2003 Feb;35(2):75-82. doi: 10.1002/ppul.10191. PMID 12526066
- [Background] Morgan WJ, Stern DA, Sherrill DL, Guerra S, Holberg CJ, Guilbert TW, Taussig LM, Wright AL, Martinez FD. Outcome of asthma and wheezing in the first 6 years of life: follow-up through adolescence. Am J Respir Crit Care Med. 2005 Nov 15;172(10):1253-8. doi: 10.1164/rccm.200504-525OC. Epub 2005 Aug 18. PMID 16109980
- [Background] Illi S, von Mutius E, Lau S, Niggemann B, Gruber C, Wahn U; Multicentre Allergy Study (MAS) group. Perennial allergen sensitisation early in life and chronic asthma in children: a birth cohort study. Lancet. 2006 Aug 26;368(9537):763-70. doi: 10.1016/S0140-6736(06)69286-6. PMID 16935687
- [Background] Zielen S, Christmann M, Kloska M, Dogan-Yildiz G, Lieb A, Rosewich M, Schubert R, Rose MA, Schulze J. Predicting short term response to anti-inflammatory therapy in young children with asthma. Curr Med Res Opin. 2010 Feb;26(2):483-92. doi: 10.1185/03007990903485148. PMID 20001651
- [Background] Beydon N, Davis SD, Lombardi E, Allen JL, Arets HG, Aurora P, Bisgaard H, Davis GM, Ducharme FM, Eigen H, Gappa M, Gaultier C, Gustafsson PM, Hall GL, Hantos Z, Healy MJ, Jones MH, Klug B, Lodrup Carlsen KC, McKenzie SA, Marchal F, Mayer OH, Merkus PJ, Morris MG, Oostveen E, Pillow JJ, Seddon PC, Silverman M, Sly PD, Stocks J, Tepper RS, Vilozni D, Wilson NM; American Thoracic Society/European Respiratory Society Working Group on Infant and Young Children Pulmonary Function Testing. An official American Thoracic Society/European Respiratory Society statement: pulmonary function testing in preschool children. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1304-45. doi: 10.1164/rccm.200605-642ST. No abstract available. PMID 17545458
- [Background] Christmann M, Erffa Sv, Rosewich M, Rose MA, Schulze J, Zielen S. [The repeatability of forced expiratory manoeuvres in 4- to 6-year-old children with intermittent bronchial asthma in healthy and in exacerbated status]. Pneumologie. 2010 Dec;64(12):745-51. doi: 10.1055/s-0030-1255625. Epub 2010 Aug 23. German. PMID 20734282
- [Background] Schulze J, Rosewich M, Riemer C, Dressler M, Rose MA, Zielen S. Methacholine challenge--comparison of an ATS protocol to a new rapid single concentration technique. Respir Med. 2009 Dec;103(12):1898-903. doi: 10.1016/j.rmed.2009.06.007. Epub 2009 Jul 10. PMID 19596563